CLINICAL TRIAL: NCT06366997
Title: Multicenter Clinical Research for Diagnosis of Epithelial Ovarian Cancer Using OCS Test
Brief Title: Diagnosis of Epithelial Ovarian Cancer Using Ovarian Cancer Score (OCS) Test
Status: Completed | Type: Observational
Sponsor: Chongqing University Cancer Hospital (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The First Affiliated Hospital of Zhengzhou University (Other); 3D Medicines Corporation (Unknown)
Responsible Party: Sponsor
Other Study IDs: CQGOG0207
Record Dates: First submitted 2024-03-13; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Epithelial Ovarian Cancer; Adnexal Mass
Keywords: early diagnosis; ovarian cancer; OCS test
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Disease; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is designed to confirm the performance of the 3D Medicines Corporation OCS test in diagnosis of epithelial ovarian cancer in patients with adnexal mass. To this end, blood samples from female patients with adnexal mass required surgical resection from four centers are obtained and analysis in the study.

ELIGIBILITY:
Inclusion Criteria:

* a) ≥ 18 years of age;
* b) Patients with adnexal masses;
* c) Sign the informed consent form;
* d) Adnexal mass that requires excision;

Exclusion Criteria:

* a) history of chemoradiotherapy;
* b) history of malignancy;
* c) pregnancy;
* d) Adnexal mass not require surgical excision;
* e) The adnexal mass has been diagnosed as malignant before surgery, and the number of cases enrolled in a single institution exceeds 50;
* f) Blood CA125 value greater than 1000 U/ml at initial treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adnexal masses (i.e., lumps near the uterus or in or around the ovaries, fallopian tubes, or surrounding connecting tissues) are common and are often detected by primary care providers and gynecologists. Adnexal masses are seen in up to 35% of premenopausal women and 17% of postmenopausal women and can occur throughout a woman's life. Although the majority of these masses are benign, they must be evaluated to rule out the possibility of malignant ovarian cancer. Ovarian cancer is one of the most aggressive gynecologic tumors worldwide, with over 31,4000 new cases diagnosed and 21,3000 deaths each year1,2. Ovarian cancer is the most lethal gynecologic malignancy with an overall 5-year survival rate of 45%.
Sampling Method: Probability Sample
Enrollment: 1352 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
the Performance of Discrimination of Benign Disease and Malignant tumors by the OCS Value. | Data analysis would be completed in three months after all data were collected.
  Evaluation of the performance of the OCS value in discriminating between benign and malignant tumors. Serum was collected before surgery. The serum OCS value was calculated with the serum level of extracellular vesicle biomarkers using a preset formula. The unit for each EV biomarker in the formula was as follows: Carbohydrate antigen 125 (CA125, U/ml), Human Epididymis Protein (HE4, pmol/L) and Complement Component 5a (5a, ng/ml). The OCS value was a numerical value witout units. The OCS value above the preset cut-off (0.506) value indicated maligant tumor, otherwise the adnexal mass was benign. The concordance between the pathological results (gold standard) and the results predicted by the OCS value was compared.

CONTACTS AND LOCATIONS:
Overall Officials: Qi Zhou, Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- No.181, Hanyulu Road, Shapingba District, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Wang H, Zhu J, Zou D, Rao Q, Han L, Lu H, Wang J, Liu L, Ma L, Sun L, Yi L, Feng W, Zhang Y, Du Y, Yang M, Feng Y, Zhang D, Lin Z, Zhou Q. Multicenter study of ovarian cancer score for diagnosing ovarian cancer. Gynecol Oncol. 2025 Feb;193:58-64. doi: 10.1016/j.ygyno.2024.12.017. Epub 2025 Jan 9. PMID 39793443